CLINICAL TRIAL: NCT03734835
Title: The Effect of Supplementation of Flaxseed, Hesperidin, Flaxseed and Hesperidin Together in Metabolic Syndrome and Its Components: A Randomized, Controlled Study
Brief Title: The Effect of Supplementation of Flaxseed, Hesperidin, Flaxseed and Hesperidin Together in Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13678
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Hesperidin; Linseed Oil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- hesperidin and flaxseed (Active Comparator): 1000 mg hesperidin as two capsules and 30 grams flaxseed
  Interventions: Dietary Supplement: hesperidin and flaxseed
- control (Placebo Comparator): no supplementation
  Interventions: Other: control
- flaxseed (Active Comparator): 30 grams flaxseed
  Interventions: Dietary Supplement: flaxseed
- hesperidin (Active Comparator): 1000 mg hesperidin as two capsules
  Interventions: Dietary Supplement: hesperidin

INTERVENTIONS:
Dietary Supplement: hesperidin — 1000 mg hesperidin as two capsules
  Arms: hesperidin
Dietary Supplement: hesperidin and flaxseed — 1000 mg hesperidin as two capsules and 30 grams flaxseed
  Arms: hesperidin and flaxseed
Dietary Supplement: flaxseed — 30 grams flaxseed
  Arms: flaxseed
Other: control — no supplementation
  Arms: control

SUMMARY:
To study the effects of Hesperidin, flaxseed and both together in patients with metabolic syndrome, 100 patients will be randomly allocated to one of following four groups: control group, hesperidin group (2 capsules Hesperidin), flaxseed group (30 gram flaxseed) or flaxseed-hesperidin group (2 capsules Hesperidin and 30 gram flaxseed) for 12 weeks; both groups will be advised to adherence the investigators' diet and exercise program too. At the first and the end of the intervention, metabolic factors will be assessed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 70 years
* having 3 of 5 of high blood sugar, hypertension, high TG, high waist circumference, low HD

Exclusion Criteria:

* pregnancy or lactation
* history of Cardiovascular disease, Pulmonary disease, Renal disease & Celiac disease; Cirrhosis
* Following a program to lose weight in recent 3 mo

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic syndrome: Number of participants with treated metabolic syndrome | 12 weeks
  Number of participants with treated metabolic syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehran, Iran (the Islamic Republic Of), Iran